CLINICAL TRIAL: NCT02090322
Title: Study of no Inferiority Between Two Doses (0.500mg and 0.625mg) of Bevacizumab Intravitreal in the Treatment of Retinopathy of Prematurity Type 1
Brief Title: Bevacizumab 0.500MG Intravitreal There Isn't Lower Than 0.625MG in the Treatment of ROP Type 1
Acronym: Bevacizumab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Martha Giselda Rangel Charqueño, Dra.Martha Giselda Rangel Charqueño, Universidad Autonoma de San Luis Potosí
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 72-12
Record Dates: First submitted 2014-02-20; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; Bevacizumab; No inferiority
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab; Angiogenesis Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): The treatment for Retinopathy of prematurity is Intravitreal bevacizumab. We want to compare two dosages (0.500 and 0.625mg) and demonstrate that 0.500mg there isn't lower in efficacy than 0.625mg.
  When the baby have the diagnosis or Retinopathy of prematurity we are going to inyect the eye that have te problem, then we are going to explore until this illness disappear. It is only one intervention
  Interventions: Procedure: Injection of bevacizumab intravitreal (Avastin)

INTERVENTIONS:
Procedure: Injection of bevacizumab intravitreal (Avastin) — The treatment of Retinopathy of prematurity is with bevacizumab intravitreal for resolution of the illness.
  When there is a Retinopathy of prematurity type 1, is the indication for the infection
  Other Names: Antiangiogenic; Avastin

SUMMARY:
The Retinopathy of Prematurity (ROP) is a Retina's pathology only of the premature baby, it's characterized for proliferation of vascular tissue that grow in the limit between the vascular retina and the avascular retina. The altered regulation of Vascular Endothelial Grow Factor (VEGF) has been proposed as one of the principal factor in the pathogenesis of the ROP.

The ROP is classified for: location (zones I,II,III), extension (hours 1 to 12) and for stages (1,2,3,4a,4b,5) and features of the vessels (normal, pre-plus and plus).

With the diagnosis of ROP type 1(ROP zone I any stage with plus, zone I stage 3 without plus, zone II stage 2 y 3 with plus) the treatment is begun and ROP type 2 is maintained in observation.

The altered regulation of Vascular Endothelial Grow Factor (VEGF) has been proposed as one of the principal factors in the pathogenesis of ROP.

DETAILED DESCRIPTION:
ustification: Before the treatment was with Cryotherapy and the standard gold is the laser, however the retina tissue is destroyed, and there is loss of visual field and as this procedure has need to be with general anesthesia, there may be trans and post surgical complications. Currently the intravitreal antiangiogenics are been employed (that inhibit the VEGF), specially the Bevacizumab, it's a quickly procedure with topic anesthesia and low price, with a good results.

It's known that intravitreal bevacizumab arrives blood and there aren't reports of secondary efects in this moment, however, we want demonstrate that for the weight and volume of the premature baby's eye, we need a low dosis and then we will have less sistemic effect.

HYPOTHESIS:The injection of 0.500 mg of Bevacizumab intravitreal it isnt lower that 0.625 mg of Bevacizumab intravitreal for the regression of ROP type 1 OBJECTIVE: Demonstrate that 0.500mg of Bevacizumab intravitreal isn't inferior that 0.625mg in the resolution of ROP type 1.

METHODOLOGY: No inferiority study. ECCA. We are going to include premature patients prematures with less of 32SDG and/or 1500g and less of 36SDG with factors risk. They are going to be examined in the week fourth, with de diagnosis for ROP type 1, we are going to inject intravitreal Bevacizumab, with the dosis randomized (0.500mg and 0.625mg) and they are going to be examined another time at first week, two weeks, first month, and for the second to sixth month after the treatment, for warrant la resolution of ROP. The size simple is 30 patients for group (Dosis A and Dosis B).

We are going to describe the date of the infection, and the age of the baby when the bevacizumab was inyected. When the ROP have been in regression, we are going to describe the date, and finally we are going to describe the age is going to be the baby she the ROP have been in regression.

It is going to be important determine the concept of exit and failure. And finally demonstrate if the two dosage have a good result

ELIGIBILITY:
Inclusion Criteria:

* Prematurity, low weight, oxygen, retinopathy of prematurity type 1

Exclusion Criteria:

* Retinopathy of prematurity type 2, retinopathy of prematurity stage 4 or 5

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Regression of Retinopathy of prematurity | 4 months
  Injection of bevacizumab and regression of this

CONTACTS AND LOCATIONS:
Overall Officials: Rangel Ch Martha, Speciality, Principal Investigator — Universidad Autonoma de San Luis Potosí
Locations (2):
- Mexico (2):
  - Hospital Central Dr. "IMP", Mexico, San Luis Potosí
  - Hospital Central Dr."IMP", Mexico, San Luis Potosí